CLINICAL TRIAL: NCT06090500
Title: Effect of Submucosal Cryotherapy Compared to Steroidal and Non-Steroidal Anti-Inflammatory Drugs Injection on Postoperative Endodontic Pain
Brief Title: Effect of Submucosal Cryotherapy on Postoperative Endodontic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mai Shalabi, Teaching Assistant in the department of endodontics faculty of dentistry ASU, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FDASU 1234
Record Dates: First submitted 2023-10-10; First posted 2023-10-19 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Post-endodontic Pain
MeSH Terms: interventions — Cryotherapy; Diclofenac; dexamethasone 21-phosphate

STUDY DESIGN:
Intervention Model Description: submucosal injection of cold saline 2 to 5 degrees celsius for cryotherapy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Submucosal Cryotherapy (Experimental): preoperative submucosal infiltration injection of (2.5C-5C) cold saline
  Interventions: Procedure: Cryotherapy
- Submucosal NSAIDs (Active Comparator): preoperative submucosal infiltration injection of Diclofenac sodium
  Interventions: Procedure: Diclofenac sodium
- Submucosal corticosteroids (Active Comparator): preoperative submucosal infiltration injection of dexamethasone
  Interventions: Procedure: Dexamethasone sodium phosphate
- Control (No Intervention): no preoperative injection apart from the normal anaesthetic routine

INTERVENTIONS:
Procedure: Cryotherapy — preoperative submucosal infiltration injection of cold saline solution (2-5 degrees Celsius)
  Arms: Submucosal Cryotherapy
Procedure: Diclofenac sodium — preoperative submucosal infiltration injection of Diclofenac sodium (25mg/ml)
  Arms: Submucosal NSAIDs
Procedure: Dexamethasone sodium phosphate — preoperative submucosal infiltration injection of dexamethasone sodium phosphate (4mg/ml)
  Arms: Submucosal corticosteroids

SUMMARY:
The goal of this clinical trial is to compare submucosal Cryotherapy with different anti-inflammatory drugs in the reduction of post-endodontic pain in upper premolars with symptomatic irreversible pulpitis.

The main question it aims to answer is:

Is there is a difference in post-endodontic pain intensity following submucosal cryotherapy or anti-inflammatory drugs injection in patients with symptomatic irreversible pulpitis? Participants will undergo root canal treatment preceded by preoperative injection of cold saline (cryotherapy) or preoperative injection of anti-inflammatory drugs Researchers will compare [Cryotherapy, Non steroidal anti-inflammatory drugs, steroids and no intervention] to see the intensity of post-endodontic pain.

DETAILED DESCRIPTION:
The study will be conducted on 52 maxillary premolar teeth; with 13 maxillary premolars in each group (n=13). An independent individual withholding the random allocation sequence, will preoperatively inform a second individual responsible for injection, about the solution required to be injected according to the patient number in the preformed randomized sequence. Triple blinding will be maintained in this study as the operator, the patients and the outcome assessor will not be aware of their group/used sub-mucosal injection.

Group I: (Diclofenac Sodium) submucosal infiltration injection of 1 ml diclofenac sodium (25mg/ml) after the normal local anaesthetic routine.

Group II: (Dexamethasone) Submucosal infiltration injection of 1 ml dexamethasone sodium phosphate (4mg/ml) after the normal local anaesthetic routine..

Group III: (Cryotherapy) Submucosal infiltration injection of 1 mL cryo-treated saline maintained at a temperature of 2 to 5°C after the normal local anaesthetic routine..

Group IV: (Negative control) Patients received no injection apart from the normal local anaesthetic routine.

Procedural steps:

1. Vitality will be assessed using cold tests before the procedure is carried out. Besides, mobility, palpation, and percussion tests will be done to assess periapical health. In order to ensure that the cold and electrical pulp tests are working, and a response is elicited, both tests will be carried out on patients not included in the study.
2. All the patients will receive local anesthesia: 4% Articaine hydrochloride with 1:100,000 epinephrine.
3. In group I submucosal infiltration injection of 1 ml diclofenac sodium (25mg/ml) will be given in the depth of the vestibule 5 minutes after local anesthetic injection.
4. In group II submucosal infiltration injection of 1 ml dexamethasone sodium phosphate (4mg/ml) will be given in the depth of the vestibule 5 minutes after local anesthetic injection.
5. In group III submucosal infiltration injection of 1 mL (2 to 5°C) cold saline will be given in the depth of the vestibule 5 minutes after local anesthetic injection.
6. In group IV regular endodontic treatment starts 5 minutes after local anesthetic injection.
7. Each tooth will be isolated using a rubber dam, and the access cavity will be prepared using a tapered diamond stone with rounded end under copious water cooling.
8. After removal of coronal pulp tissues using a sterile excavator, the working length will be determined with stainless steel hand K-files size #10 and the use of an apex locator and confirmed using intraoral periapical radiographs.
9. Hand instrumentation to 15-size K files.
10. All the canals will be prepared using M-Pro Gold rotary files till the master apical file.
11. Apical patency will be maintained throughout the shaping procedure using the #10 file between each instrument.
12. All the canals will be irrigated with 10 mL of 5.25% NaOCl between each file during the whole preparation procedure.
13. After completion of cleaning and shaping canals will be dried using appropriate size paper points and obturated using gutta-percha with cold lateral technique, then restored by temporary restoration

ELIGIBILITY:
Inclusion Criteria:

* Egyptian healthy both gender patients (Category: American Society of Anesthesiologists ASA class I)
* Patients age (18- 50) years old.
* Maxillary premolar teeth diagnosed with symptomatic irreversible pulpitis.
* No clinical or radiographic evidence of periapical nor periodontal pathosis.
* Compliant patient.

Exclusion Criteria:

* The vulnerable group; prisoners, pregnant females, mentally ill, severe systemic diseases, psychological diseases, TMJ problems.
* Analgesics or anti-inflammatory drugs taken within 24 h before the intervention.
* Over instrumentation during treatment.
* Long-term use of corticosteroids.
* Access revealing necrotic tooth indicating a false positive diagnosis.
* Sensitivity to any of the pharmaceuticals intended to be used in this study.
* Intra operative complications such as canal calcification, or loss of apical Patency.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
the level of post-endodontic pain | 6 hours after completion of endodontic treatment
  Evaluation of the pain intensity using the Numeric Rating Scale. The Numeric Rating Scale measures pain intensity. Numeric Rating Scale consists of scores ranged from 0-10,with lowest 0 as lowest score representing ('no pain') and 10 as highest score representing ('pain as bad as it could possibly be)
the level of post-endodontic pain | 24 hours after completion of endodontic treatment
  Evaluation of the pain intensity using the Numeric Rating Scale. The Numeric Rating Scale measures pain intensity. Numeric Rating Scale consists of scores ranged from 0-10,with lowest 0 as lowest score representing ('no pain') and 10 as highest score representing ('pain as bad as it could possibly be)
the level of post-endodontic pain | 48 hours after completion of endodontic treatment
  Evaluation of the pain intensity using the Numeric Rating Scale. The Numeric Rating Scale measures pain intensity. Numeric Rating Scale consists of scores ranged from 0-10,with lowest 0 as lowest score representing ('no pain') and 10 as highest score representing ('pain as bad as it could possibly be)
the level of post-endodontic pain | 72 hours after completion of endodontic treatment
  Evaluation of the pain intensity using the Numeric Rating Scale. The Numeric Rating Scale measures pain intensity. Numeric Rating Scale consists of scores ranged from 0-10,with lowest 0 as lowest score representing ('no pain') and 10 as highest score representing ('pain as bad as it could possibly be)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt